CLINICAL TRIAL: NCT01129336
Title: A Multicenter, Open-label, Randomized Trial to Evaluate the Anti-cancer Effects of Zoledronic Acid and Circulating Tumor Cell Measurements in Patients With HER2-negative Metastatic Breast Cancer Without Bone Metastasis
Brief Title: Effect of Zoledronic Acid as Anti-Cancer Treatment in Metastatic Breast Cancer Patients
Acronym: MACS1295
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EUS147
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: First or Second Line HER2-negative Breast Cancer; Metastatic Disease Without Bone Metastasis
Keywords: HER2-negative; HER2; Metastatic breast cancer; First Line breast cancer; Second Line breast cancer; Breast cancer; Metastatic; Stage IV breast cancer; Progression free survival; PFS; Circulating Tumor Cells; CTCs; Zoledronic acid; HER2-negative metastatic breast cancer patients without bone metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplastic Cells, Circulating | interventions — Zoledronic Acid; Diphosphonates; Standard of Care

ARMS (2):
- Patients without bone metastases (Experimental): Patients with no bone metastasis were randomized into a 1:1 ratio to standard therapy plus zoledronic acid 4mg IV Zoledronic acid administration monthly during Months 1-18.
  Interventions: Drug: Zoledronic acid
- Patients with bone metastases (Experimental): Patients with bone metastasis received standard therapy + zoledronic acid for 18 months (discontinued upon disease progression/secondary malignancy)
  Interventions: Drug: Standard Therapy

INTERVENTIONS:
Drug: Zoledronic acid — Patients with no bone metastasis (n=150) will receive Standard therapy plus Zoledronic acid administration 4 mg IV monthly during Months 1-18.
  Other Names: Zometa; bisphosphonates; CZOL446E
  Arms: Patients without bone metastases
Drug: Standard Therapy — Standard Therapy, including chemotherapy and hormonal therapy, was determined at the discretion of the investigator.
  Arms: Patients with bone metastases

SUMMARY:
This study will evaluate zoledronic acid's anti-cancer effects and Circulating Tumor Cell (CTCs) measurements in patients with HER2-negative metastatic breast cancer without bone metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female patients (age ≥18 years)
* HER2-negative metastatic breast cancer (stage IV)
* Patients will be receiving chemotherapy or hormonal therapy
* Patients with no bone metastasis and ≤1 prior treatments for metastatic breast cancer. Patients with newly diagnosed metastatic breast cancer may have received adjuvant or neoadjuvant chemotherapy as long as treatment was completed ≥12 months prior to relapse.
* Asymptomatic brain metastasis is permitted if all of the following criteria are met:

  1. no sign of clinical progression or known progression of brain metastasis
  2. off steroids for at least 2 weeks prior to study enrollment
* Stable renal function: two serum creatinine determinations of <3 mg/dL, obtained no less than 7 days apart (one value may be obtained within 6 weeks prior to Screening; the second must be obtained during Screening)
* ECOG performance status of 0 or 1
* Life expectancy of ≥ 6 months
* Negative serum pregnancy test
* Ability and willingness to comply with all study requirements

Exclusion Criteria:

* Known hypersensitivity to zoledronic acid or other bisphosphonates
* Patients with history of another malignancy within the last two years prior to study enrollment, except cured basal cell carcinoma of the skin or excised carcinoma in site of the cervix
* Use of concurrent investigational agents is prohibited. Prior use of investigational agents is permitted if discontinued ≥30 days prior to Screening.
* No prior therapy with an antiresorptive agent
* Patients with active brain metastases or meningeal metastases
* Current or recent (in the six months prior to initial study drug treatment) severe cardiovascular disease (defined as uncontrolled congestive heart failure), hypertension refractory to treatment, or poorly controlled Type I/II diabetes mellitus
* Current active dental problems including dental abscess or infection of the jawbone (maxilla or mandible) or a current or prior diagnosis of osteonecrosis of the jaw
* Patients who have received radiotherapy ≤ 4 weeks prior to study enrollment or who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to study enrollment is allowed
* Patients who have undergone major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) ≤ 4 weeks prior to study enrollment or who have not recovered from side effects of such therapy
* Diminished renal capacity: calculated creatinine clearance (CrCl) <30 mL/min (based on Cockcroft-Gault formula)
* Corrected (i.e., adjusted for serum albumin) serum calcium of <8.0 mg/dL (2.00 mmol/L) or ≥ 12 mg/dL (3.00 mmol/L)
* Pregnant or breast-feeding females
* Women of child-bearing potential who are not willing/able to use effective methods of birth control (e.g., abstinence, oral contraceptives or implants, IUD, vaginal diaphragm or sponge, or condom with spermicide)
* History of non-compliance to medical regimens and/or patients who are considered unreliable
* History of bone metabolism diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- United States (33):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Clopton Clinic, Jonesboro, Arkansas
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Kaiser Permanente Medical Group Kaiser Permanente - Hawaii, Anaheim, California
  - Wilshire Oncology Medical Group, La Verne, California
  - Loma Linda University Loma Linda Cancer Center, Loma Linda, California
  - Hematology and Medical Oncology, Waterbury, Connecticut
  - Florida Cancer Specialists DeptofFloridaCancerSpecialists, Fort Myers, Florida
  - Lakeland Regional Cancer Center Dept. of Lakeland Regional, Lakeland, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - Kootenai Medical Center Kootenai Medical Center, Coeur d'Alene, Idaho
  - Oncology Specialists, SC Lutheran General Cancer Instit, Park Ridge, Illinois
  - Cancer Center of Kansas, Witchita, Kansas
  - Park Nicollet Institute Dept. of Park Nicollet, Saint Louis Park, Minnesota
  - St. John's Mercy Medical Center St. John's Mercy Med Ctr, St Louis, Missouri
  - Hematology Oncology Centers of the Northern Rockies Hema Onc Ctr N. Rockies (4, Billings, Montana
  - Southeast Nebraska Oncology Cancer Center, Lincoln, Nebraska
  - Reno Oncology Consultants, Reno, Nevada
  - Somerset Hematology Oncology Associates Somerset Hema Oncol Assoc (2), Somerset, New Jersey
  - Cooper Cancer Center, Voorhees Township, New Jersey
  - NYU Langone Arena Oncology, Lake Success, New York
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Piedmont Hematology and Oncology Associates Piedmont Hem/Onc Assoc (2), Winston-Salem, North Carolina
  - Hematology Oncology Center, Inc., Elyria, Ohio
  - Milton S Hershey Medical Center Hershey Medical Center (4), Hershey, Pennsylvania
  - Berks Hematology Oncology, West Reading, Pennsylvania
  - Abington Hematology Oncology Associates, Inc, Willow Grove, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Oncology and Hematology, PA South Texas Oncology (2), San Antonio, Texas
  - East Texas Medical Center Cancer Institute Tyler Hem/Onc (3), Tyler, Texas
  - Medical Oncology & Hematology Associates of Northern VA Med. Onc&Hem Assoc. of No.VA, Reston, Virginia
  - Northwest Medical Specialties, Tacoma, Washington

REFERENCES:
- See also: Related Info — http://www.NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 patients were screened. 44 patients received treatment.
Period: Overall Study
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases
Started | 15 | 29
Completed Treatment | 1 | 3
Completed | 3 (Completed indicates Completed Study as per protocol.) | 13 (Completed indicates Completed Study as per protocol.)
Not Completed | 12 | 16
Not completed — Protocol Violation | 1 | 0
Not completed — Disease Progression | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Missing Study Completion Status | 2 | 3
Not completed — Death | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases | Total
Number analyzed (Participants) | 15 | 29 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.48 (12.293) | 59.47 (14.535) | 57.43 (13.965)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 29 | 44
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (target or non-target) must have exhibited a reduction in short axis to < 10 mm. Partial Response (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD): at least 20% increase in sum of diameters of target lesions taking as reference the smallest sum on study accompanied by an absolute increase of at least 5 mm or appearance of one or more new lesions. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum diameters. PFS is time from enrollment to date of first documented disease progression or death due to any cause. A participant is considered to be censored when data on time to event is missing due to a subject being lost to follow-up or non-occurrence of the outcome event before the completion of the trial.
Time Frame: up to 18 months
Population: All Enrolled Patients population, which included all enrolled patients regardless of whether they received study drug.
Measure: Number; unit: Participants
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases
Number analyzed (Participants) | 15 | 29
Participants
  Event | 9 | 19
  Censor | 6 | 10

2. Secondary Outcome: Percentage of Patients With Circulating Tumor Cell Levels of at Least 5 Per 7.5 mL of Peripheral Blood by Month
Description: Circulating tumor cells (CTCs) have been associated with poor patient prognosis and outcomes in patients receiving treatment for MBC. CTCs have been evaluated as a potential biomarker for predicting treatment effects and overall survival. Baseline was defined as the last predose measurement for patients who received any study drug and as the later of the screening visit or Visit 2 value for patients who did not receive the study drug. Percentage was calculated as the number of patients with CTC ≥5/7.5 mL against the number of patients with nonmissing CTC values (represented as 'n' in the categories).
Time Frame: Baseline, Month 1, 2, 4, 6, 9 and 18
Population: All Enrolled Patients population, which included all enrolled patients regardless of whether they received study drug. "n" in each category represents the number of patients with non-missing CTC values.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases
Number analyzed (Participants) | 15 | 29
Percentage of Participants
  Baseline (n=15,28) | 26.7 [7.8 to 55.1] | 57.1 [37.2 to 75.5]
  Month 1 (n=8,0) | 12.5 [0.3 to 52.7] | NA [NA to NA] — No patient analyzed in this arm for month 1.
  Month 2 (n=12,24) | 8.3 [0.2 to 38.5] | 25.0 [9.8 to 46.7]
  Month 4 (n=8,20) | 0 [0 to 0] | 15.0 [3.2 to 37.9]
  Month 6 (n=7,19) | 0 [0 to 0] | 15.8 [3.4 to 39.6]
  Month 9 (n=2,14) | 0 [0 to 0] | 35.7 [12.8 to 64.9]
  Month 18 (n=2,1) | 0 [0 to 0] | 100.0 [0 to 100]

3. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from the date of enrollment to the date of first documented disease progression or death due to metastatic breast cancer.
Time Frame: up to 18 months
Population: All Enrolled Patients population, which included all enrolled patients regardless of whether they received study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases
Number analyzed (Participants) | 15 | 29
Days | 190 [118 to 478] | 297 [221 to 373]

4. Secondary Outcome: Change From Baseline in Urine NTX by Month
Description: NTX= N-telopeptide of type 1 collagen (nmol bce/mmol [nanomoles of bone collagen equivalents per millimole of creatinine]). Baseline was defined as the last predose measurement for patients who received any study drug and as the later of the screening visit or visit 2 value for patients who did not receive study drug.
Time Frame: Baseline, Month 2, Month 4
Population: All Enrolled Patients population, which included all enrolled patients regardless of whether they received study drug.
Measure: Mean (Standard Deviation); unit: nmol bce/mmol
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases
Number analyzed (Participants) | 15 | 29
nmol bce/mmol
  Change from baseline at Month 2 | -5.25 (22.5555) | -27.619 (23.3955)
  Change from baseline at Month 4 | -4.750 (18.7521) | -23.476 (26.3526)

ADVERSE EVENTS:
Arm/Group | Patients Without Bone Metastases | Patients With Bone Metastases
Serious Adverse Events (participants affected / at risk) | 2/15 | 7/29
Other Adverse Events (participants affected / at risk) | 13/15 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Without Bone Metastases (N=15) | Patients With Bone Metastases (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Without Bone Metastases (N=15) | Patients With Bone Metastases (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 4
Deafness (Ear and labyrinth disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 8
Oedema mouth (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 4
Fatigue (General disorders) | 4 | 18
Generalised oedema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 3 | 3
Pain (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 5
Jaundice (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 0 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 6
Haemoglobin decreased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 2
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Sinus headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 4
Sleep disorder (Psychiatric disorders) | 1 | 0
Bladder irritation (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 5
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 3
Lymphoedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.